CLINICAL TRIAL: NCT04676477
Title: A Phase 1 Open-Label Study of HER3-DXd (Patritumab Deruxtecan; U3-1402) in Combination With Osimertinib in Subjects With Locally Advanced or Metastatic EGFR-mutated Non-Small Cell Lung Cancer (NSCLC)
Brief Title: HER3-DXd (Patritumab Deruxtecan; U3-1402) in Combination With Osimertinib in Subjects With Locally Advanced or Metastatic EGFR-mutated Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: U31402-A-U103; 2020-003064-87 (EudraCT Number)
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Advanced Non-small Cell Lung Cancer; Inoperable Non-small Cell Lung Cancer; HER3-DXd (Patritumab Deruxtecan; U3-1402); Unresectable; Epidermal growth factor receptor; Metastatic; EGFR; Osimertinib; HER3
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — patritumab deruxtecan; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation: HER3-DXd + osimertinib (Experimental): Participants in the Dose Escalation phase will receive HER3-DXd IV Q3W + osimertinib PO once daily. The dose of HER3-DXd in the first cohort will be 3.2 mg/kg Q3W. The dose of osimertinib in the first cohort will be 80 mg PO once daily.
  Interventions: Drug: HER3-DXd; Drug: Osimertinib
- Second-line Dose Expansion: HER3-DXd + osimertinib (RCD) (Experimental): Participants in the Second-line Dose Expansion phase will be randomized to receive HER3-DXd + osimertinib at the RCD
  Interventions: Drug: HER3-DXd; Drug: Osimertinib
- Second-line Dose Expansion: HER3-DXd (Experimental): Participants in the Second-line Dose Expansion phase will be randomized to receive HER3-DXd 5.6 mg/kg IV Q3W
  Interventions: Drug: HER3-DXd
- First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 3; RCD) (Experimental): If the RCD includes an osimertinib dose of 80 mg PO once daily, then participants will receive treatment with HER3-DXd and osimertinib at the RCD
  Interventions: Drug: HER3-DXd; Drug: Osimertinib
- First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 4a) (Experimental): Participants in the First-line Dose Expansion phase will be randomized to receive HER3-DXd 5.6 mg/kg IV Q3W and osimertinib dose of 80 mg PO once daily.
  Interventions: Drug: HER3-DXd; Drug: Osimertinib
- First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 4b) (Experimental): Participants in the First-line Dose Expansion phase will be randomized to receive HER3-DXd 4.8 mg/kg IV Q3W and osimertinib dose of 80 mg PO once daily.
  Interventions: Drug: HER3-DXd; Drug: Osimertinib

INTERVENTIONS:
Drug: HER3-DXd — Intravenous infusion at a starting dose of 3.2 mg/kg Q3W
  Other Names: U3-1402; Patritumab deruxtecan
  Arms: Dose Escalation: HER3-DXd + osimertinib
Drug: HER3-DXd — Intravenous infusion at RCD 1 (and at RCD 2 if two provisional RCDs are selected in dose escalation)
  Other Names: U3-1402; Patritumab deruxtecan
  Arms: First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 3; RCD); Second-line Dose Expansion: HER3-DXd + osimertinib (RCD)
Drug: Osimertinib — Oral administration at 40 mg or 80 mg once daily
  Arms: Dose Escalation: HER3-DXd + osimertinib
Drug: Osimertinib — Oral administration at RCD 1 (and at RCD 2 if two provisional RCDs are selected in dose escalation)
  Arms: First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 3; RCD); Second-line Dose Expansion: HER3-DXd + osimertinib (RCD)
Drug: HER3-DXd — Intravenous infusion 5.6 mg/kg Q3W
  Other Names: U3-1402; Patritumab deruxtecan
  Arms: First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 4a); Second-line Dose Expansion: HER3-DXd
Drug: HER3-DXd — Intravenous infusion 4.8 mg/kg Q3W
  Other Names: U3-1402; Patritumab deruxtecan
  Arms: First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 4b)
Drug: Osimertinib — Oral administration at 80 mg once daily
  Arms: First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 4a); First-line Dose Expansion: HER3-DXd + osimertinib (Cohort 4b)

SUMMARY:
This study includes a Dose Escalation Part to identify the recommended combination dose (RCD) and a Dose Expansion Part to further evaluate efficacy and safety.

The primary objectives:

Dose Escalation: To assess the safety and tolerability of HER3-DXd (patritumab deruxtecan; U3-1402) and osimertinib in subjects with locally advanced or metastatic non-small cell lung cancer (NSCLC) with an EGFR exon 19 deletion or L858R mutation with tumor progression after treatment with osimertinib, and to determine the recommended combination dose (RCD).

Second-Line Dose Expansion Arm 1 and Arm 1b: To assess the preliminary antitumor activity of HER3-DXd and osimertinib in subjects with locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation with tumor progression after treatment with osimertinib. Note: One or both of the study arms may open with one or two distinct dosing schedules.

Second-Line Dose Expansion Arm 2: To assess the preliminary antitumor activity of HER3-DXd monotherapy in subjects with locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation with tumor progression after treatment with osimertinib.

First-Line Dose Expansion Cohorts 3, 4a, and 4b: To assess the preliminary antitumor activity of HER3-DXd and osimertinib in subjects with locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation without prior systemic treatment for locally advanced or metastatic disease.

DETAILED DESCRIPTION:
Dose Escalation:

Population includes subjects with locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation with tumor progression after treatment with osimertinib. The starting combination dose regimen is HER3-DXd 3.2 mg/kg IV every 21 days (Q3W) and osimertinib 80 mg orally (PO) once daily. At least 3 to 6 subjects will be enrolled in each cohort.

Dose Expansion: Two subject populations will be evaluated in the Dose Expansion Part:

* Second-Line: Subjects with locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation with tumor progression after treatment with osimertinib
* First-Line: Subjects with locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation, and without prior systemic therapy for advanced or metastatic disease. Note: The first line expansion will only be initiated if the RCD includes osimertinib 80 mg PO once daily.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Specific to Dose Escalation and Second-line Dose Expansion:

* Documentation of EGFR exon 19 deletion or L858R mutation detected from tumor tissue
* Must have received osimertinib for locally advanced or metastatic disease at a dose of 80 mg once daily (QD) for at least 6 weeks and must not miss more than two doses during the 2 weeks prior to the first day of study treatment (Cycle 1, Day 1)
* Must not have received any other prior systemic cancer therapies in the locally advanced/metastatic setting
* Has documentation of radiological disease progression following first-line treatment with osimertinib in the locally advanced or metastatic setting

Inclusion Criteria Specific to First-line Dose Expansion:

* The tumor tissue harbors one of the 2 common EGFR mutations occurring in NSCLC known to be associated with EGFR-TKI sensitivity (exon 19 deletion or L858R) as assessed by Clinical Laboratory Improvement Amendments (CLIA)-certified (United States [US] sites), accredited (outside of the US), local laboratory or central laboratory. Only tissue-based testing will be accepted.
* Participants must have previously untreated locally advanced or metastatic NSCLC and must be eligible to receive first-line treatment with osimertinib, according to the judgment of the investigator. Prior adjuvant or neo-adjuvant therapy (chemotherapy, radiotherapy, investigational agents; except with osimertinib) is permitted.

All Participants:

Participants must meet all criteria to be eligible for inclusion in this study:

* Histologically or cytologically documented locally advanced or metastatic NSCLC not amenable to curative surgery or radiation.
* At least 1 measurable lesion as assessed by Investigator as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
* Tissue requirements

  * For Dose Escalation (all cohorts): provide an optional pre-treatment tumor tissue of sufficient quantity, as defined in the laboratory manual. The optional pre-treatment tumor tissue can be provided as either:

    * Pre-treatment tumor biopsy from at least 1 lesion not previously irradiated and amenable to core biopsy OR
    * Archival tissue collected from a biopsy performed prior to signing of the tissue consent, and since progression while on treatment with the most recent cancer therapy
  * For First-line Dose Expansion (Cohorts 3, 4a, and 4b): provide an optional pre-treatment and optional on-treatment tumor tissues of sufficient quantity, as defined in the laboratory manual. The optional pre-treatment tumor tissue can be provided as either:

    * Pre-treatment tumor biopsy from at least 1 lesion not previously irradiated and amenable to core biopsy OR
    * Archival tissue collected from a biopsy performed at the time of initial diagnosis or later
  * For Second-line Dose Expansion (Arm 1, Arm 2, and Arm 1b): provide a required pre-treatment and required on-treatment tumor tissues of sufficient quantity, as defined in the laboratory manual. The required pre-treatment tumor tissue can be provided as either:

    * Pre-treatment tumor biopsy from at least 1 lesion not previously irradiated and amenable to core biopsy OR
    * Archival tissue collected from a biopsy performed prior to signing of the tissue consent, and since progression while on treatment with the most recent cancer therapy regimen

      * Note: For all participants who consent to a pre-treatment biopsy, in order to ensure an adequate amount of tissue is available, a core needle biopsy is required.
* Has adequate bone marrow reserve and organ function based on local laboratory data within 14 days prior to Cycle 1, Day 1 (Dose Escalation and First-line Dose Expansion) or within 14 days prior to randomization (Second-line Dose Expansion):

  * Platelet count: ≥100 000/mm^3 or ≥100 × 10^9/L (platelet transfusions are not allowed within 14 days prior to the assessment of platelets during the screening period in order to meet the study inclusion criterion)
  * Hemoglobin: ≥9.0 g/dL (transfusion of red blood cells and/or growth factor support is not allowed within 14 days prior to the assessment of hemoglobin during the screening period in order to meet the study inclusion criterion)
  * Absolute neutrophil count (ANC): 1500/mm^3 or ≥1.5 × 10^9/L (granulocyte colony stimulating factor support is not allowed within 14 days prior to the assessment of ANC during the screening period in order to meet the study inclusion criterion)
  * Creatinine clearance (CrCl): CrCl ≥30 mL/min as calculated using the Cockcroft-Gault equation or measured CrCl
  * Aspartate aminotransferase/ alanine aminotransferase: ≤3 × ULN (if liver metastases are present, ≤5 × ULN)
  * Total bilirubin: ≤1.5 × ULN if no liver metastases (<3 × ULN in the presence of documented Gilbert's syndrome [unconjugated hyperbilirubinemia] or liver metastases)
  * Serum albumin: ≥2.5 g/dL
  * Alkaline phosphatase (ALP) and Gamma-glutamyl transferase (GGT): ≤2.5 × ULN of both ALP and GGT
  * Prothrombin time (PT) or PT-international normalized ratio (INR) and Activated partial thromboplastin time (aPTT) / Partial thromboplastin time (PTT): ≤1.5 × ULN, except for subjects on coumarin-derivative anticoagulants or other similar anticoagulant therapy, who must have PT-INR within therapeutic range as deemed appropriate by the Investigator.

Exclusion Criteria:

* Any previously documented histologic or cytologic evidence of small cell OR combined small cell/non-small cell disease
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroid therapy, has current ILD, or is suspected to have such disease by imaging during screening.
* Clinically severe pulmonary compromise (based on Investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

  * Any underlying pulmonary disorder (eg, pulmonary emboli within three months of the study enrollment or randomization, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion);
  * Any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (eg, rheumatoid arthritis, Sjogren's syndrome, sarcoidosis); OR prior complete pneumonectomy.
* Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to Cycle 1, Day 1. Participants who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study.
* Evidence of any leptomeningeal disease.
* Has spinal cord compression or clinically active central nervous system metastases, defined as symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Participants with clinically inactive brain metastases may be included in the study. Participants with treated brain metastases who are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study, but must have a stable neurologic status for at least 4 weeks prior to Cycle 1, Day 1. Participants with asymptomatic brain metastases and treated with anticonvulsants as prophylaxis are able to enroll following a 14-day washout period. Note: A CT or MRI scan of the brain at baseline is required for all participants.
* Inadequate washout period prior to Cycle 1, Day 1 defined as:

  * Whole brain radiation therapy <28 days or stereotactic brain radiation therapy <7 days;
  * Any systemic anticancer therapy (excluding osimertinib in all Dose Escalation Cohorts and in Second-line Dose Expansion [Arm 1, Arm 2, and Arm 1b]), including investigational agents, <14 days or 5 half-lives, whichever is longer
  * Immune checkpoint inhibitor therapy ≤21 days
  * Major surgery (excluding placement of vascular access) <4 weeks
  * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation < 28 days or palliative radiation therapy <7 days
  * Chloroquine or hydroxychloroquine ≤14 days
  * Medications or herbal supplemented known to be strong inducers of cytochrome P450 (CYP) 3A4 <21 days.
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, Grade ≤1 or baseline. Subjects with chronic Grade 2 toxicities may be eligible per the discretion of the Investigator after consultation with the Sponsor Medical Monitor or designee.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow osimertinib, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
* Has any primary malignancy other than locally advanced or metastatic NSCLC within 3 years prior to Cycle 1, Day 1 (Dose Escalation and First-line Dose Expansion) or within 3 years prior to randomization (Second-Line Dose Expansion), except adequately resected non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated.
* Uncontrolled or significant cardiovascular disease prior to Cycle 1, Day 1 including:

  * Mean corrected QT interval using Fridericia's formula (QTcF) interval of >450 ms in 3 successive central screening measurements
  * Left ventricular ejection fraction (LVEF) ≤50% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan
  * Resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg
  * Myocardial infarction within 6 months
  * New York Heart Association (NYHA) Classes 2 to 4 congestive heart failure within 28 days
  * Uncontrolled angina pectoris within 6 months
  * Has cardiac arrhythmia requiring antiarrhythmic treatment
  * Complete left or right bundle branch block within 6 months
  * History of second- or third-degree heart block or PR interval >250 ms within 6 months
  * History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes
  * Has any factors that increase the risk of corrected QT (QTc) prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives, or any concomitant medication known to prolong the QT interval
* Has clinically significant corneal disease
* Any evidence of severe or uncontrolled diseases including active bleeding diatheses, active infection, psychiatric illness/social situations, geographical factors, substance abuse, or other factors which in the Investigator's opinion makes it undesirable for the subject to participate in the study or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required.
* Has a known human immunodeficiency virus (HIV) infection that is not well controlled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Incidence of Dose-limiting Toxicities (DLT), Treatment-emergent Adverse Events (TEAE), Serious Adverse Events (SAE), Adverse Events of Special Interest (AESI) | From signing of informed consent form up to 40 days (+7 days) after the last dose of study drugs, up to approximately 9 months
  A DLT is defined as any TEAE not attributable to disease or disease-related processes that occurs during the DLT evaluation period and is ≥Grade 3, as defined in the protocol. A TEAE is defined as an adverse event (AE) with a start or worsening date during the on-treatment period. A serious AE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event, or may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes noted. AESIs will also be assessed. AEs will be coded using MedDRA and graded using NCI-CTCAE v5.0.
Second-line Dose Expansion and First-line Dose Expansion: Objective Response Rate (ORR) | From start of study treatment until date of documented disease progression or other protocol-defined reason for discontinuation from the study (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 18 months
  ORR is defined as the proportion of participants who achieved a best overall response of confirmed complete response (CR) or confirmed partial response (PR) as assessed by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors version (RECIST) v1.1.

SECONDARY OUTCOMES:
Dose Escalation: Objective Response Rate (ORR) | From start of treatment until date of disease progression or other reason for discontinuation (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 9 months (Dose Escalation) and 18 months (Dose Expansion)
  ORR is defined as the proportion of participants who achieved a best overall response of confirmed CR or confirmed PR as assessed by BICR and Investigator per RECIST v1.1.
Second-line Dose Expansion and First-line Dose Expansion: Objective Response Rate (ORR) | From start of study treatment until the date of documented disease progression or other protocol-defined reason for discontinuation from the study (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 18 months
  ORR is defined as the proportion of participants who achieved a best overall response of confirmed CR or PR as assessed by Investigator per RECIST v1.1.
Dose Escalation, Second-line Dose Expansion, and First-Line Dose Expansion: Duration of Response (DoR) | From start of treatment until date of disease progression or other reason for discontinuation (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 9 months (Dose Escalation) and 18 months (Dose Expansion)
  DOR is defined as the time from the date of the first documentation of response (confirmed CR or confirmed PR) to the date of the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first. DoR as assessed by BICR and Investigator per RECIST v1.1
Second-line Dose Expansion: Clinical Benefit Rate (CBR) | From start of treatment until date of disease progression or other reason for discontinuation (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 9 months (Dose Escalation) and 18 months (Dose Expansion)
  CBR is defined as the proportion of participants who have a confirmed best overall response of CR, PR, or SD that lasts for at least 180 days as assessed by BICR and Investigator per RECIST v1.1.
Dose Escalation, Second-line Dose Expansion, and First-line Dose Expansion: Disease Control Rate (DCR) | From start of treatment until date of disease progression or other reason for discontinuation (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 9 months (Dose Escalation) and 18 months (Dose Expansion)
  DCR is defined as the proportion of participants who achieved a best overall response of confirmed CR, confirmed PR, or stable disease (SD) as assessed by BICR and by Investigator per RECIST v1.1.
Dose Escalation, Second-line Dose Expansion, and First-line Dose Expansion: Time to Response (TTR) | From start of treatment until date of disease progression or other reason for discontinuation (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 9 months (Dose Escalation) and 18 months (Dose Expansion)
  TTR is defined as the time from the start of study treatment to the date of the first documentation of response (confirmed CR or confirmed PR) in responding participants as assessed by BICR and by Investigator per RECIST v1.1.
Dose Escalation, Second-line Dose Expansion, and First-line Dose Expansion: Progression-free Survival (PFS) | From start of treatment until date of disease progression or other reason for discontinuation (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 9 months (Dose Escalation) and 18 months (Dose Expansion)
  PFS is defined as the time from the start of study treatment to the date of the first documentation of objective PD as assessed by BICR and by Investigator per RECIST v1.1. or death due to any cause, whichever occurs first
Dose Escalation, Second-line Dose Expansion, and First-line Dose Expansion: Overall Survival (OS) | From start of treatment until date of disease progression or other reason for discontinuation (e.g, withdrawal of consent, lost to follow-up), whichever occurs first, up to approximately 9 months (Dose Escalation) and 18 months (Dose Expansion)
  OS is defined as the time from the start of study treatment to the date of death due to any cause.
Second-line Dose Expansion and First-line Dose Expansion: Incidence of Treatment-emergent Adverse Events (TEAE), Serious Adverse Events (SAE), Adverse Events of Special Interest (AESI) | From signing of informed consent form up to 40 (+7 days) days after the last dose of study drugs, up to approximately 18 months
  A TEAE is defined as an adverse event (AE) with a start or worsening date during the on-treatment period. A serious AE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event, or may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes noted. AESIs will also be assessed. Adverse events will be coded using MedDRA and will be graded using NCI-CTCAE v5.0.
Dose Escalation, Second-line Dose Expansion, and First-line Dose Expansion: Proportion of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) and Proportion of Participants Who Have Treatment-emergent ADA | From the start of study treatment until the end of treatment or study discontinuation (whichever occurs first), up to approximately 9 months (Dose Escalation) and 18 months (Dose Expansion)
  The immunogenicity of HER3-DXd will be assessed.
Dose Escalation, Second-line Dose Expansion, and First-line Dose Expansion: Pharmacokinetic Parameter Maximum Concentration (Cmax) | HER3-DXd: Cycles 1 and 3, Day 1 pre- and postdose, 4 hours (h), Days 8 and 15; Cycle 2, Day 1 pre- and postdose; Cycles 4, 6, 8, Day 1 pre- and postdose; Osimertinib: Cycles 1, 2, and 3, Day 1 pre- and postdose, 4 h (each cycle is 21 days)
  Cmax will be assessed for HER3-DXd (anti-HER3-ac-DXd, total anti-HER3 antibody LC-MS and DXd), osimertinib (except for Second-line Dose Expansion Arm 2), and AZ5104 (active metabolite of osimertinib; except for Second-line Dose Expansion Arm 2).
Dose Escalation, Second-line Dose Expansion, and First-line Dose Expansion: Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) | HER3-DXd: Cycles 1 and 3, Day 1 pre- and postdose, 4 hours (h), Days 8 and 15; Cycle 2, Day 1 pre- and postdose; Cycles 4, 6, 8, Day 1 pre- and postdose; Osimertinib: Cycles 1, 2, and 3, Day 1 pre- and postdose, 4 h (each cycle is 21 days)
  Tmax will be assessed for HER3-DXd (anti-HER3-ac-DXd, total anti-HER3 antibody LC-MS and DXd), osimertinib (except for Second-line Dose Expansion Arm 2), and AZ5104 (active metabolite of osimertinib; except for Second-line Dose Expansion Arm 2).
Dose Escalation, Second-line Dose Expansion, and First-line Dose Expansion: Pharmacokinetic Parameter Area Under the Concentration-Time Curve (AUC) | HER3-DXd: Cycles 1 and 3, Day 1 pre- and postdose, 4 hours (h), Days 8 and 15; Cycle 2, Day 1 pre- and postdose; Cycles 4, 6, 8, Day 1 pre- and postdose; Osimertinib: Cycles 1, 2, and 3, Day 1 pre- and postdose, 4 h (each cycle is 21 days)
  AUC up to the last quantifiable time (AUClast) and AUC during dosing interval (AUCtau) will be assessed for HER3-DXd (anti-HER3-ac-DXd, total anti-HER3 antibody LC-MS and DXd), osimertinib (except for Second-line Dose Expansion Arm 2), and AZ5104 (active metabolite of osimertinib; except for Second-line Dose Expansion Arm 2).

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (31):
- United States (13):
  - UCLA, Santa Monica, California
  - Yale University School of Medicine - Yale-New Haven Hospital, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Japan (10):
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Okayama University Hospital, Okayama, Okayama-ken
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni-shi, Yamaguchi
  - Kindai University Hospital, Ōsaka-sayama
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital of JFCR, Tokyo
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (4):
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/